CLINICAL TRIAL: NCT02254538
Title: A Double-blind (at Each Dose Level), Randomised, Placebo-controlled Single Increasing Dose Safety, Tolerability and Preliminary Pharmacokinetics Study in Healthy Male Volunteers After Oral Administration of BILR 355 BS Solved in PEG 400 (Dosage: 1 - 200 mg)
Brief Title: A Safety, Tolerability and Preliminary Pharmacokinetics of BILR 355 BS Single-rising Dose Study in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1188.1
Record Dates: First submitted 2014-09-29; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — polyethylene glycol 400

ARMS (2):
- BILR 355 BS (Experimental): escalating doses
  Interventions: Drug: BILR 355 BS; Drug: PEG 400
- Placebo (Placebo Comparator)
  Interventions: Drug: PEG 400

INTERVENTIONS:
Drug: BILR 355 BS
  Arms: BILR 355 BS
Drug: PEG 400

SUMMARY:
Assessment of safety, tolerability and preliminary pharmacokinetics in healthy male volunteers after oral administration of BILR 355 BS

ELIGIBILITY:
Inclusion Criteria:

All participants in the study should be healthy males, ranging from 21 to 50 years of age and their body mass index (BMI) be within 18.5 to 29.9 kg/m2 (BMI calculation: weight in kilograms divided by the square of height in meters).

In accordance with Good clinical practice (GCP) and the local legislation all volunteers will have given their written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (≤ two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (≥ 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the clinically accepted reference range
* Excessive physical activities within the last week before the trial or during the trial

Following exclusion criteria are of special interest for this study:

- Erythema, exanthema and comparable skin alterations

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2002-05; Primary Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinically significant changes in vital functions | Up to 10 days after drug administration
Number of participants with abnormal findings in ECG (electrocardiogram) | Up to 10 days after drug administration
Number of participants with abnormal findings in skin inspections | Up to 10 days after drug administration
Number of participants with abnormal neurological finding | Up to 10 days after drug administration
Number of participants with abnormal changes in laboratory parameters | Up to 10 days after drug administration
Number of participants with positive faecal occult blood testing | Up to 10 days after drug administration
Number of participants with adverse events | Up to 10 days after drug administration

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Up to 144 hours after drug administration
Time to attain maximum plasma concentration (tmax) | Up to 144 hours after drug administration
Area under the concentration-time curve of the analyte in plasma from zero time to infinity (AUC0-∞) | Up to 144 hours after drug administration
Terminal half life (t½) | Up to 144 hours after drug administration
Apparent clearance of the analyte in plasma following extravascular administration (CL/F) | Up to 144 hours after drug administration
Total mean residence time (MRTtot) | Up to 144 hours after drug administration
Apparent volume of distribution during the terminal elimination phase (Vz/F) | Up to 144 hours after drug administration
Renal clearance of the analyte (CLR) | Up to 72 hours after drug administration
Amount of drug excreted in the urine (Ae) | Up to 72 hours after drug administration
Area under the concentration-time curve of the analyte in plasma from zero time to the time of the last quantifiable drug concentration (AUC0-tz) | Up to 144 hours after drug administration